CLINICAL TRIAL: NCT02834143
Title: Evaluation of Diagnostic Criteria for Chronic Critical Limb Ischemia
Acronym: CRIMI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CRIMI
Record Dates: First submitted 2016-07-07; First posted 2016-07-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-07

CONDITIONS: Stroke
Keywords: vascular; Limb Ischemia
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — The is no intervention. This study is a descriptive one

SUMMARY:
Chronic critical limb ischemia (CCI) is the most severe clinical form of occlusive arterial disease. Its prognosis is terrible, mortality estimated at 50% in five years. However there are no recent epidemiological data on morbidity and mortality of critical ischemia. Moreover, the diagnostic criteria of the ICC associate clinical and hemodynamic criteria and are not subject to a clear consensus.

Investigators propose to evaluate the validated diagnostic criteria (TASC VALMI, European working group) in a population of severe ischemia in patients in order to offer relevant simple and reproducible criteria. Secondly Investigators propose to monitor the medium and long term evolution of these patients ICC defined to clarify the prognosis.

diagnostic criteria of the different societies:

* TASC: Transatlantic criteria: very characteristic pain, wound optional, variable hemodynamic criteria as the presence of a wound or not
* VALMI: French criteria derived vascular medical college: characteristic pain, sore, hemodynamic reproducible, reliable criteria
* European working group: European definition of criteria, including a characteristic pain, requires no wound, different hemodynamic criteria of 2 others.

DETAILED DESCRIPTION:
Main objective / secondary:

* Main objective: Evaluation of diagnostic criteria for chronic critical limb ischemia
* Secondary objectives:

  * Evaluation of the quality of life,
  * Evaluation of the need for psychological counseling a patient at the stage of chronic critical limb ischemia,
  * Evaluation of the interest of a specific bioassay

Development of the study:

The offer document and the non-opposition of the patient will be collected on the first day of hospitalization, quality of life questionnaires will also be distributed at the beginning of hospitalization.

Clinical data will be collected during hospitalization of the patient, respecting their anonymity, only the place of birth shall be retained in terms of data that distinguish patients.

During the consultation of control, a half months post-hospitalization, diagnostic criteria will be reviewed and the quality of life (using the same questionnaire) and the need or not for psychological help (oral question).

The doctor will be called between 3 and 6 months following hospitalization to assess her patient monitoring criteria, rhythm monitoring, the psychological impact of the disease on the patient seen by the physician, assessment loss of independence due to illness.

The number of hospitalizations for chronic critical ischemia of six months shall be obtained.

Methodology :

Design: Prospective, mono centric, non-interventional (observational) consecutive patients attending the service Vascular Medicine.

Study duration: 6 months: about 150 to 180 patients included in the study, about 50 have clinical chronic critical limb ischemia criteria.

ELIGIBILITY:
Inclusion Criteria:

* All patients suffering from peripheral arterial disease of the lower limbs hospitalized in vascular medicine department of GHPSJ and having a life expectancy greater than one year.

Exclusion Criteria:

* demented patient psychological condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients suffering from peripheral arterial disease of the lower limbs hospitalized in vascular medicine department of GHPSJ (Groupe Hospitalier Paris Saint Joseph) and having a life expectancy greater than one year.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2015-01-14 (Actual); Study Completion 2015-06-14 (Actual)

PRIMARY OUTCOMES:
Assessent of change of The Trans-Atlantic Inter-Society Consensus Document on Management of Peripheral Arterial Disease (TASC) | Day 1, then Day 45 after hospitalization
Assessent of change of VALMI (French criteria derived vascular medical college) | Day 1, then Day 45 after hospitalization
  French criteria derived vascular medical college: characteristic pain, sore, reproducible hemodynamic criteria, reliable
Assessent of change of the European working group criteria | Day 1, then Day 45 after hospitalization
  European definition of criteria, including a characteristic pain, requires no wound, different haemodynamic criteria 2 others.

SECONDARY OUTCOMES:
Assessent of quality of life | Day 1, then Day 45 after hospitalization
  Quality of Life questionnaire validated by the French Society of Angiology (SF 12)
Evaluation of the need for psychological counseling | Day 1, then Day 45 after hospitalization
  Evaluation of the need of the patient for psychological counseling at the stage of chronic critical limb ischemia: questions posed orally directly to the patient "do you feel the need for psychological counseling? "(When viewing control, a month and a half after hospitalization)
  Possible answers are : yes or no
Evaluation of the interest of a specific bioassay | Day 1, then Day 45 after hospitalization
  Evaluation of the interest of a specific bioassay: no additional assay carried out for the study, only biologies prescribed as part of its usual management will be carried out
  Possible answers are : yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Michon Pasturel Ulrique, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided